CLINICAL TRIAL: NCT07279025
Title: Symptom Evaluation and Quantification for Unified Outcomes and Individualized Assessment
Brief Title: Validate the Temporal Stability and Responsiveness of AI-COA® for Depression and Anxiety
Acronym: SEQUOIA-2
Status: Not yet recruiting | Type: Observational
Sponsor: Deliberate Solutions Inc. (Industry)
Collaborators: Baylor College of Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: SEQUOIA-2
Record Dates: First submitted 2025-12-07; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Depression Disorders; Anxiety Disorders
Keywords: depression assessment; anxiety assessment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — audiovideo recordings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the reliability and responsiveness of the AI-COA®, a digital tool designed to assess the severity of depression and anxiety. The study compares the tool's performance against standard clinician ratings over 12 weeks to determine its consistency and sensitivity to symptom changes.

DETAILED DESCRIPTION:
The SEQUOIA-2 study evaluates the effectiveness of Artificial Intelligence (AI) in measuring depression and anxiety severity in adults. Investigators from Deliberate Solutions, Inc. and Baylor College of Medicine are conducting this study to determine whether AI can provide reliable clinical assessments of mood and anxiety disorders. The study compares the tool's performance against standard clinician ratings over a 12-week period to determine its consistency and sensitivity to symptom changes.

In clinical trials for new depression and anxiety treatments, human clinicians typically conduct interviews to evaluate participants' symptoms. These assessments are critical but may vary based on the clinician's experience or interview style, potentially affecting the reliability of research findings.

To address this challenge, the study team developed an AI-based Clinical Outcome Assessment tool, called AI-COA®, which analyzes video interviews to measure symptoms of depression and anxiety consistently and objectively. AI-COA® has been accepted by the U.S. Food and Drug Administration (FDA) into the Innovative Science and Technology Approaches for New Drugs (ISTAND) pilot program.

The primary objectives of the SEQUOIA-2 study are to confirm test-retest reliability (whether the tool produces consistent scores when symptoms are stable) and sensitivity to change (whether the tool accurately detects changes in symptom severity over time compared to standard clinical scales).

Participants will undergo a series of remote, video-recorded clinical interviews conducted by trained clinicians. The study uses standard clinical outcome assessments as reference standards. The recorded data will be processed by the tool to assess its agreement with human raters. Participants will also complete questionnaires about their symptoms and perform brief tasks.

The development and validation of reliable, AI-driven assessment tools through this study aim to enhance the accuracy of mental health evaluations, potentially improving the testing and approval processes for new treatments targeting depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* 18 to 65 years of age.
* HAM-D 17 > 10
* Starting, or has started, a new treatment for depression or anxiety within 2-3 weeks of enrollment
* Access to a laptop or other computer with a well functioning microphone and webcam, and a stable Internet connection
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Resides in the United States at the time of consent and during completion of study

Exclusion Criteria:

* Any cognitive impairment that limits ability to provide informed consent or authorization
* Vulnerable or protected populations (e.g. prisoners)
* Impairment that would prevent participants from completing an online survey and/or engaging in clinician assessment interviews (e.g., visual impairment, motor impairment, hearing impairment)
* Acute intoxication at the time of the assessments
* Concurrent medication/treatment:

  * Receiving any fast-acting treatment for depression or anxiety (e.g. ketamine, psychedelics, deep brain stimulation, etc.) in between initial baseline assessment (A1) and Restest (A2) , or in between Follow up assessment (B1) and Retest (B2)
  * Anxiolytics: Use of benzodiazepines or other anxiety-reducing medications that could affect speech or motor activity, within the past 4 weeks.
  * Antipsychotics and Mood Stabilizers: Medications that can alter cognitive and motor functions, within the past 6 weeks.
  * Stimulants: Use of medications like methylphenidate or amphetamines that affect energy levels and behavior, within the past 2 weeks
  * Epilepsy medication: seizure activity or medication side effects that may alter behavior, within the past 4 weeks.
* Any history or evidence of any of the following conditions:

  * Neurodevelopmental, Neurocognitive, Neurodegenerative or movement disorders including, but not limited to:
  * Tourette's syndrome
  * Multiple Sclerosis
  * Amyotrophic Lateral Sclerosis
  * Parkinson's Disease
  * Stroke
  * Traumatic Brain Injury
  * Facial paralysis.
* Conditions with vocal cord impact:

  * Vocal cord injury or cerebrovascular accident or head trauma with residual dysarthria in the past year
  * Disorders that may impact vocal cords such as acute or chronic laryngitis, vocal cord paresis or paralysis, or spasmodic dysphonia
  * Past or active heavy smokers (an average of >20 cigarettes per day)
* Schizophrenia Spectrum and Other Psychotic Disorders:

  * Individuals with a current or past diagnosis of Schizophrenia, Schizoaffective Disorder, or other psychotic disorders, including Delusional Disorder and Brief Psychotic Disorder.
  * Current hypomanic episode as defined by DSM-5 criteria. This includes those with Bipolar I Disorder, Bipolar II Disorder, or Cyclothymic Disorder who are not in a stable mood state at the time of assessment.
  * Chronic Pain Conditions: Such as fibromyalgia, which may affect facial expressions and vocal tone.
  * Prosthetic Facial Devices: Could affect facial recognition algorithms. Cosmetic Procedures: Such as Botox injections or facelifts that can impact facial expressions.
  * Dental Work: Major procedures that might affect speech.
* Participants who have previously participated in another research project by Deliberate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with MDD or MDE
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
HAM-D ICC | Between Test and Retest (within 2 days)
  Concordance of HAM-D score between model and human raters

SECONDARY OUTCOMES:
MADRS ICC | Between Test and Retest (within 2 days)
  Concordance of MADRS score between model and human raters
HAM-A ICC | Between Test and Retest (within 2 days)
  Concordance of HAM-A score between model and human raters

CONTACTS AND LOCATIONS:
Overall Officials: Marc Aafjes, Principal Investigator — Deliberate Solutions Inc.
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No